CLINICAL TRIAL: NCT04609735
Title: Manual Therapy, Exercise and Ultrasound Vs. Manual Therapy, Exercise, Ultrasound and Electric Dry Needling for Patients With Medial Epicondylalgia
Brief Title: Manual Therapy, Exercise and US Vs. Manual Therapy, Exercise and US for Medial Epicondylalgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alabama Physical Therapy & Acupuncture (Other)
Collaborators: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, James Dunning, DPT, MSc, FAAOMPT, Director, American Academy of Manipulative Therapy, Alabama Physical Therapy & Acupuncture
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAMT50
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Epicondylalgia
MeSH Terms: interventions — Musculoskeletal Manipulations; Exercise; High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Electric DN, Manual therapy, exercise and US (Experimental): Dry needling, manual therapy, exercise and ultrasound
  Interventions: Other: Electric Dry Needling, Manual Therapy, Exercise and Ultrasound
- Active comparator: Manual therapy, exercise and ultrasound (Active Comparator): Active comparator: Manual therapy, exercise and ultrasound
  Interventions: Other: Manual Therapy, Exercise and Ultrasound

INTERVENTIONS:
Other: Electric Dry Needling, Manual Therapy, Exercise and Ultrasound — Electric Dry Needling, Manual Therapy, Exercise and Ultrasound
  Arms: Experimental: Electric DN, Manual therapy, exercise and US
Other: Manual Therapy, Exercise and Ultrasound — Electric Dry Needling, Manual Therapy, Exercise and Ultrasound vs. Manual Therapy, Exercise and Ultrasound
  Arms: Active comparator: Manual therapy, exercise and ultrasound

SUMMARY:
The purpose of this research is to compare two different approaches for treating patients with medial epicondylalgia: manual therapy, exercise and ultrasound and manual therapy, exercise, ultrasound and electric dry needling. Physical therapists commonly use all of these techniques to treat medial epicondylalgia. This study is attempting to find out if one treatment strategy is more effective than the other.

DETAILED DESCRIPTION:
Patients with medial epicondylalgia will be randomized to receive 8 treatments (2 treatments per week) over 4 weeks (8 treatments max) of either: 1. manual therapy, exercise and ultrasound or 2. manual therapy, exercise, ultrasound and electric dry needling

ELIGIBILITY:
Inclusion Criteria:

1. Adult between18 and 60 years old that is able to speak English.
2. Report of at least 6 weeks of elbow (i.e. medial epicondyle) and ventral forearm pain, consistent with medial epicondylalgia.
3. Patient has not had physical therapy, massage therapy, chiropractic treatment or injections for elbow pain in the last 6 months.
4. Diagnosis of medial epicondylalgia, defined as the following:(Walz, 2010; Shin, 2019)

   1. Tenderness is elicited by palpation of the insertion of the flexor-pronator mass (5-10 mm distal and anterior to the middle aspect of the medial epicondyle)
   2. Pain is exacerbated by resisted wrist flexion and forearm pronation at an angle of 90°

Exclusion Criteria:

1. Report of red flags to manual physical therapy to include: severe hypertension, infection, uncontrolled diabetes, peripheral neuropathy, heart disease, stroke, chronic ischemia, edema, severe varicosities, tumor, metabolic disease, prolonged steroid use, fracture, RA, osteoporosis, severe vascular disease, malignancy, etc.
2. Report of Previous surgery of the elbow, history of elbow dislocation, elbow fracture and/or tendon rupture.
3. History of or presentation consistent with osteochondritis dissecans, osteoarthrosis, MCL injury (i.e. Pain with valgus stress or positive "milking test" - pulling on the thumb with the elbow in flexion and the forearm in supination), flexor-pronator strain, and ulnar neuropathy (i.e. Positive Tinel sign - distal pain and tingling during direct compression of the nerve at the elbow).
4. Report of systemic neurological disorders and/or neurological deficits to include the following: a. Nerve root compression (muscle weakness involving a major muscle group of the upper extremity, diminished upper extremity deep tendon reflex, or diminished or absent sensation to pinprick in any upper extremity dermatome) b. Cervical or thoracic spinal stenosis (exhibited by bilateral upper extremity symptoms) c. Central nervous system involvement (hyperreflexia, sensory disturbances in the hand, intrinsic muscle wasting of the hands, unsteadiness during walking, nystagmus, loss of visual acuity, impaired sensation of the face, altered taste, the presence of pathological reflexes) d. History of whiplash or T-spine injury injury within the previous 6 weeks 5. History of surgery to the head/neck/T-spine or affected upper extremity.

6. Psychiatric disorders or cognitively impaired 7. Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-10-31 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in elbow pain intensity (NPRS) | Baseline, 1-week, 4-weeks, 3-months
  Numeric Pain Rating Score. Higher scores mean greater pain

SECONDARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand | Baseline, 1-week, 4-weeks, 3-months
  The DASH is measured on a 0-100 scale. Greater scores indicate increased disability.
Change in Global rating of change score | 4-weeks, 3-months
  Global rating of change - Scale = -7 to 7. Greater numbers represent a perceived improvement of symptoms, while lesser scores indicate a perceived worsening of symptoms
Change in Medication Intake (Frequency of Medication Intake in last week) | Baseline, 3-months
  Frequency of medication intake in last week

CONTACTS AND LOCATIONS:
Overall Officials: James Dunning, DPT PhD, Principal Investigator — American Academy of Manipulative Therapy
Locations (1):
- Mallers and Swoverland Orthopedic PT, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided